CLINICAL TRIAL: NCT00319683
Title: A Phase 1/2 Study in Subjects With Locally Advanced, Recurrent, or Metastatic Hepatocellular Carcinoma, Evaluating the Safety, and Anti-Tumor Activity of ADH300004 (Eniluracil) With Escalating Doses of 5 Fluorouracil Administered Orally Once Weekly for 3 Weeks Out of Every 4 (Adherex Protocol Number AHX-03-103)
Brief Title: A Study of ADH300004 and 5-Fluorouracil in Locally Advanced, Recurrent, or Metastatic Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Adherex Technologies, Inc. (Industry)
Responsible Party: Clinical Study Manager, Adherex Technologies
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHX-03-103
Expanded Access: Available
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Cancer; Tumors; Neoplasms; Anticarcinogenic Agents; Antineoplastic Agents; Dihydrouracil Dehydrogenase (NADP)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms | interventions — eniluracil

INTERVENTIONS:
Drug: ADH300004

SUMMARY:
5-fluorouracil (5-FU), one of the most actively investigated anti-cancer drugs, is rapidly inactivated by the enzyme dihydropyrimidine dehydrogenase (DPD). ADH300004 blocks DPD. This study will test the safety and effects of oral ADH300004 14 hours prior to oral 5-FU in subjects with locally advanced, recurrent, or metastatic hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* In the Phase I portion, Asian subjects that are > or = to 18 years of age
* In the Phase II portion, any subjects that are > or = to 18 years of age
* Non-resectable locally advanced, recurrent, or metastatic hepatocellular carcinoma (HCC) that is either histologically proven or a radiologically documented liver mass with: (alpha-fetoprotein [AFP] > 4,000 ng/mL, hepatitis B surface antigen positive or alpha-fetoprotein [AFP] > 400 ng/mL, hepatitis B surface antigen negative)
* Radiologically documented measurable disease
* Adequate performance status and organ function, as evidenced by hematologic and biochemical blood testing
* Willing to not receive fluoropyrimidine containing chemotherapy for 8 weeks after the last dose of ADH300004 in this study

Exclusion Criteria:

* Chemotherapy, radiotherapy, or any other investigational drug within 28 days prior to study entry
* No more than 1 previous treatment with systemic chemotherapy (chemotherapy administered as part of a chemo-embolization procedure is not considered systemic chemotherapy)
* Portal hypertension with bleeding esophageal or gastric varices within the past 3 months
* Ascites that is refractory to conservative management
* Inability to take oral medication
* Active peptic ulcer disease
* Known hypersensitivity to 5-FU or ADH300004
* History of primary brain tumors or brain metastases
* Previous or concurrent malignancy at another site within the last 5 years
* Stroke, major surgery, or other major tissue injury within 30 days before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Whang-Peng, MD, Principal Investigator — National Health Research Institute, Ward Veterans General Hospital
Locations (7):
- Queens Medical Center, Honolulu, Hawaii, United States
- Johns Hopkins Singapore International Medical Center, Singapore, Singapore
- Taiwan (5):
  - Chang Gung Memorial Hospital, Chiayi City
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City
  - National Health Research Institute, Ward Veterans General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

REFERENCES:
- See also: Adherex Technologies Inc. Corporate Homepage — http://www.adherex.com